CLINICAL TRIAL: NCT06985121
Title: Evaluation of the Scalp Skin Care Effects of Premium Scalp Revitalizing Essence、Premium Scalp Revitalizing Essence 2、Premium Scalp Revitalizing Essence 3
Brief Title: Scalp Care Efficacy Evaluation for Premium Scalp Revitalizing Essence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hungkuang University (Other)
Responsible Party: Principal Investigator, Tsong-Min Chang, Vice President, Hungkuang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25-016-A
Record Dates: First submitted 2025-05-20; First posted 2025-05-22 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-06

CONDITIONS: Scalp Health; Hair Condition; Hair Loss; Sebum Production; Hair and Scalp Health
Keywords: Scalp care; Hair loss; Skin texture; Sebum measurement; Scalp condition; Hair length; Hair density; Cosmetics; Product formulation; Growth factor; Centella asiatica; Extracellular vesicles
MeSH Terms: conditions — Alopecia | interventions — Insulin-Like Growth Factor I

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1: Placebo control (Placebo Comparator): Base formula without caffeine and panthenol
  Interventions: Other: Placebo control
- Group 2: Base formula only (Experimental): Base formula consisting of active ingredients caffeine and panthenol (vitamin B5).
  Interventions: Other: Base formula only
- Group 3: Base formula plus IGF-1 & FGF-7. (Experimental): Base formula plus insulin growth factor 1 (IGF-1) and fibroblast growth factor-7 (FGF-7)
  Interventions: Other: Base formula plus IGF-1 and FGF-7
- Base formula plus Centella asiatica extracellular vesicles (Experimental): Base formula plus Centella asiatica extracellular vesicles
  Interventions: Other: Base formula plus Centella asiatica extracellular vesicles
- Group 5: Base formula plus Centella asiatica extracellular vesicles, IGF-1 & FGF-7. (Experimental): Base formula plus Centella asiatica extracellular vesicles, insulin growth factor-1 (IGF-1) and fibroblast growth factor-7 (FGF-7).
  Interventions: Other: Base formula plus Centella asiatica extracellular vesicles, IGF-1 & FGF-7

INTERVENTIONS:
Other: Placebo control — Placebo control (base formula without caffeine and panthenol). Applied 1mL evenly to the scalp once daily after hair wash for 56 consecutive days.
  Arms: Group 1: Placebo control
Other: Base formula only — Base formula consisting of active ingredients caffeine and panthenol. Applied 1mL evenly to the scalp once daily after hair wash for 56 consecutive days.
  Arms: Group 2: Base formula only
Other: Base formula plus IGF-1 and FGF-7 — Base formula plus insulin growth factor 1 (IGF-1) and fibroblast growth factor-7 (FGF-7). Applied 1mL evenly to the scalp once daily after hair wash for 56 consecutive days.
  Arms: Group 3: Base formula plus IGF-1 & FGF-7.
Other: Base formula plus Centella asiatica extracellular vesicles — Base formula plus Centella asiatica extracellular vesicles. Applied 1mL evenly to the scalp once daily after hair wash for 56 consecutive days.
  Arms: Base formula plus Centella asiatica extracellular vesicles
Other: Base formula plus Centella asiatica extracellular vesicles, IGF-1 & FGF-7 — Base formula plus Centella asiatica extracellular vesicles, insulin growth factor-1 (IGF-1) and fibroblast growth factor-7 (FGF-7). Applied 1mL evenly to the scalp once daily after hair wash for 56 consecutive days.
  Arms: Group 5: Base formula plus Centella asiatica extracellular vesicles, IGF-1 & FGF-7.

SUMMARY:
The study aims to evaluate the efficacy of the Premium Scalp Revitalizing Essence on human scalp skin. A total of 60 healthy adults, aged 18 to 60, will be recruited and randomly assigned into five groups receiving different formulations. Participants will use the product once daily for 56 days, and their scalp conditions will be assessed through skin texture tests at multiple time points. Key parameters such as sebum content, overall hair loss, hair density, scalp condition, and hair length will be measured.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blinded, and placebo-controlled study to investigate the effects of Premium Scalp Revitalizing Essence on changes in the skin texture of human scalp skin.

Sixty healthy adults aged from 18 to 60 will be recruited and randomly assigned into five groups, with 12 individuals in each group. Group 1 uses Placebo (Base formula without caffeine and panthenol); Group 2 uses the Base formula (Control with caffeine and panthenol); Group 3 uses Base + IGF-1 & FGF-7; Group 4 uses Base + Centella asiatica extracellular vesicles; Group 5 uses Base + Centella Asiatica Exosome + IGF-1 & FGF-7. Before using the test product, all 60 participants undergo the first scalp skin texture test. After 14 days of using the test product, a second scalp skin texture test is conducted; after 28 days of use, a third test is performed; after 42 days of use, a fourth test is conducted; and after 56 days of use, a fifth test is carried out. The scalp skin texture tests include measurements of skin (1) sebum content, (2) overall hair loss, (3) hair density, (4) scalp condition, (5) hair length, and other parameters. The Sebumeter® SM815 probe of the MPA580 device and the ScalpX Intelligent Scalp Diagnostic System will be used to measure the parameters of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults of any gender from the age of 18 to 60 years (inclusive).
* Absence of chronic diseases, major illnesses, or allergies.
* Major illnesses include cancer, post-stroke disorders, paralysis, acute myocardial infarction, coro-nary artery bypass surgery, end-stage renal disease, and major organ transplant or hematopoietic stem cell transplant

Exclusion Criteria:

* Currently taking any medication or using any scalp care products

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Sebum Content | Assessment conducted every 14 days from Day 0 to Day 56 (including Day 0)
  Assess oil levels on the scalp at standardized scalp sites (left, right, and vertex). Measured with C+K Multi Probe Adaptor MPA580 system using the Sebumeter® SM815 probe based on the grease spot photometry method with the sebum measurement cassette tape. The change in light transmission corresponds to the amount of sebum on the tape and is displayed on a scale from 0 to 350 units.
Hair length | Assessment conducted every 14 days from Day 0 to Day 56 (including Day 0)
  Hair length (cm): Assessed with the ScalpX Intelligent Scalp Diagnostic System with digital microscopy at standardized scalp sites (left, right, and vertex).
Hair density | Assessment conducted every 14 days from Day 0 to Day 56 (including Day 0)
  Hair density (number of hairs/cm-square): Assessed with the ScalpX Intelligent Scalp Diagnostic System with digital microscopy at standardized scalp sites (left, right, and vertex).
Hair thickness | Assessment conducted every 14 days from Day 0 to Day 56 (including Day 0)
  Hair thickness (micrometers): Assessed with the ScalpX Intelligent Scalp Diagnostic System with digital microscopy at standardized scalp sites (left, right, and vertex).
Hair loss | Assessment conducted every 14 days from Day 0 to Day 56 (including Day 0)
  Hair loss: Assessed by the standardized hair combing test by counting the number of hairs shed after the participants' hair was combed over a clean surface for 60 strokes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hungkuang University, Taichung, Taiwan